CLINICAL TRIAL: NCT06159764
Title: National Registry of Cardioneuroablation in Recurrent Reflex Syncope
Acronym: CANVAS-R
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2022/62
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Syncope, Vasovagal; Bradycardia; Heart Arrest
Keywords: cardioneuroablation; vasovagal syncope; registry
MeSH Terms: conditions — Syncope, Vasovagal; Bradycardia; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cardioneuroablation: Cardioneuroablation
  Interventions: Procedure: Cardioneuroablation

INTERVENTIONS:
Procedure: Cardioneuroablation — radiofrequency ablation to destroy cardiac ganglionated plexi located in epicardial fat pads around the atrias

SUMMARY:
This registry aims to collect patient data on cardioneuroablation for vasovagal syncope from multiple centers in France. The aim is to evaluate success rates, compare techniques and help institutions set up their own cardioneuroablation program

DETAILED DESCRIPTION:
Cardioneuroablation is an emerging technique used to treat patients with vagally-mediated extrinsic bradycardia. It seems particularly efficient in patients with recurrent vasovagal syncope due to a strong cardioinhibitory effect. The procedure consists in using radiofrequency ablation to destroy cardiac ganglionated plexi located in epicardial fat pads around the atrias. Key questions concerning this procedure still remain unanswered: 1) What is the success rate of the procedure 2) Which patients will benefit from this technique? 3) Which fat pads should be targeted during the procedure? 4) What is the best way of identifying the location of these fat pads? 5) What are the long-term effects of this procedure? A multicenter registry seems ideal to try to answer these questions at minimal cost

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or more
* Recurrent vasovagal syncope (≥2 episodes during the last year) with an asystolic component (≥3 second pause) recorded during a spontaneous episode. The asystole can be related to sinus arrest or paroxysmal AV block.
* Scheduled cardioneuroablation procedure
* Estimated residual battery life ≥ 1 year.
* Patient affiliated to or beneficiary of national health security scheme.
* Patient who have received an information notice and has not objected to the use of their data in the registry.

Exclusion Criteria:

* Contraindication to anticoagulation therapy: major bleeding, risk of major bleeding, severe hepatic disease
* Contraindication to cardiac CT: contrast medium allergies
* Intracardiac thrombus
* Patient detained by judicial or administrative decision.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with vagally-mediated extrinsic bradycardia
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of vasovagal syncope | 12 months
  Number of patients with recurrence

SECONDARY OUTCOMES:
Recurrence of vasovagal syncope in different subgroups | 12 months
  Number of patients with recurrence
Efficacy of cardioneuroablation procedure | 12 months
  Number of asystolic pauses
prevalence of post-ablation pre-syncopal events | 12 months
  Number of post-ablation pre-syncopal events
correlation between ablation sites and epicardial fat pads | 12 months
  spatial correlation between ablation sites and epicardial fat pads
Quality of life of post-ablated patients (Score 1) | 12 months
  ISQoL score (Impact of syncope on quality of life) (0-55, lower scores indicate less impact of syncope on HRQoL [better]
Quality of life of post-ablated patients (Score 2) | 12 months
  SFSQ score (Syncope Functional Status HR-QoL Questionnaire) (0-100, lower scores indicate less impact of syncope [better])
Assessment of technical learning curve by centre | 12 months
  procedure time

CONTACTS AND LOCATIONS:
Overall Officials: Josselin DUCHATEAU, Principal Investigator — University Hospital, Bordeaux
Locations (14):
- France (14):
  - Hôpital Louis Pradel, Bron
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Lille, Lille
  - Hôpital de la Timone, Marseille
  - CHU de Montpellier, Montpellier
  - Clinique du Millénaire, Montpellier
  - Hôpital Pitié-Salpêtriére, Paris
  - Hôpital européen Georges Pompidou, Paris
  - Hôpital Haut-Lévèque, Pessac
  - CHR Pontchaillou, Rennes
  - Centre cardiologique du Nord, Saint-Denis
  - Institut ARNAULT TZANCK, Saint-Laurent-du-Var
  - Clinique Pasteur, Toulouse
  - CHU de Toulouse, Toulouse